CLINICAL TRIAL: NCT05810935
Title: Safety of Antibiotic Intake During Pregnancy: Results of Questionnaire of Pregnant Women in Two Arab Countries
Brief Title: Safety of Antibiotic Intake During Pregnancy
Acronym: antibiotic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Eman Ibrahim Abd Elrehim, Lecturer in Department of obstetrics and gynecology, Damietta Faculty of Medicine, Al-Azhar University, Al-Azhar University
Other Study IDs: DFM-IRB 00012367-23-03-004
Record Dates: First submitted 2023-03-29; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Infections
Keywords: antibiotics, infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study will be conducted to assess the knowledge of the pregnant females regarding safety of antibiotic intake ,also their attitude toward any prescribed antibiotics during their pregnancy .

DETAILED DESCRIPTION:
this study will be conducted on pregnant females from two Arab countries to assess their knowledge and attitude toward any prescribed antibiotics while they are pregnant .Also to assess any malpractice while their intake for any antibiotics . this study is a cross sectional study that will involve a questionnaire including the three mentioned domains .

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at any gestational age

Exclusion Criteria:

* pregnant women who refused to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: this study is an observational cross sectional study that will be conducted on pregnant female above the age of 18 years old iwith exclusion of any female with any psychological disability.
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with antibiotic-related side effects | through study completion ,an average of one year
  using a questionnaire to measure the knowledge and attitude of pregnant women toward antibiotics that were taken during pregnancy and any malpractice during its intake

IPD SHARING:
Plan to Share IPD: No